CLINICAL TRIAL: NCT06525805
Title: Readers' Attention of Shorter Versus Longer Abstracts of Systematic Reviews: A Randomized Controlled Trial
Brief Title: Readers' Attention of Shorter Versus Longer Abstracts of Systematic Reviews
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Oldenburg (Other)
Responsible Party: Principal Investigator, Jasmin Helbach, Principal Investigator, University of Oldenburg
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: UO_Abstracts_2024
Record Dates: First submitted 2024-07-18; First posted 2024-07-29 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-11

CONDITIONS: Researchers Attention

STUDY DESIGN:
Intervention Model Description: This will be a two-arm, single-blinded, superiority, parallel-group randomized controlled trial (RCT) with 1:1 allocation of intervention and control groups.
Who Masked: Participant
Masking Description: The participants will be blinded to the intervention. In the cover letter, participants will be informed that the study aims to examine the characteristics of an abstract. However, they will not be informed that the primary focus of this study is the influence of the abstract´s length. Furthermore, the participants will be not aware of the number of different abstracts that were randomly allocated.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Long Abstract (Experimental): Abstract length: 771 words
  Interventions: Other: Long Abstract
- Short Abstract (Active Comparator): Abstract length: 277 words
  Interventions: Other: Short Abstract

INTERVENTIONS:
Other: Long Abstract — The intervention and control group will be provided with a structured abstract of the review by Soderberg et al., entitled "Percutaneous nephrolithotomy vs. retrograde intrarenal surgery for renal stones". This review was published once in the Cochrane Database of Systematic Reviews and once in the journal BJU International. The length of the abstract differs significantly depending on the journal.
  The participants assigned to this study arm will be presented with the longer version published in the Cochrane Database, comprising 771 words (PMID: 37955353).
  Arms: Long Abstract
Other: Short Abstract — The participants assigned to this study arm will be presented with the shorter version published in BJU International, comprising 277 words (PMID: 37942649).
  Arms: Short Abstract

SUMMARY:
The present randomized controlled trial (RCT) was designed to investigate the perceptions of researchers on systematic review (SR) abstracts. The primary objective will be to compare readers' attention of shorter versus longer abstracts. The secondary objective will be to assess the perception of an abstract based on four indicators of a well-written abstract: (a) Informativeness, (b) Accuracy, (c) Attractiveness, and (d) Conciseness.

The study will involve researchers from all over the world who recently published an SR, regardless of their research field. To identify eligible authors, a search of MEDLINE (via PubMed) was conducted on May 5, 2024, for systematic reviews published between January 1, 2024, and March 26, 2024. A total of at least 6200 SRs will be selected from PubMed and assessed for eligibility. The corresponding author information will be extracted from all included SRs and randomized in a 1:1 ratio.

DETAILED DESCRIPTION:
This study will attempt to emulate the reading process observed in PubMed. When searching PubMed, researchers are initially presented with an overview of the references identified. After clicking on the title, the corresponding abstract appears. For full-text access, researchers must actively follow a separate link to the journal page.

In this RCT, participants will be randomly assigned in a 1:1 ratio to two groups (those receiving a long abstract vs. those receiving a short abstract). Both groups receive the same cover letter by e-mail explaining the purpose of the study, the use of the data, measures to ensure anonymity of participation, and a link for participation.

The link will direct participants to SoSci Survey, an online survey tool. Those in the group receiving the long abstract will see an abstract with a length of 771 words (PMID: 37955353). Those in the group receiving the short abstract will see an abstract with a length of 277 words (PMID: 37942649). Both abstracts are structured and pertain to the same review entitled "Percutaneous nephrolithotomy vs. retrograde intrarenal surgery for renal stones". This review was published once in the Cochrane Database of Systematic Reviews and once in the journal BJU International.

The design of the abstract presented is similar to that of PubMed, but no title or authors will be indicated. After reading the abstract, participants must actively click the "Continue" button to proceed with the survey.

ELIGIBILITY:
The corresponding authors of systematic reviews that were indexed in PubMed between January 1, 2024, and March 26, 2024, and for which an English abstract is available will be included. These include authors of all types of SR, with the majority likely representing SRs on effectiveness. Authors of other types of evidence syntheses (e.g. scoping reviews, methodological papers), editorials, protocols, corrections, retractions, erratums, or summaries of SRs will be excluded.

For identifying the systematic reviews from which the corresponding authors will be contacted we will use the following eligibility criteria.

Inclusion Criteria:

* Systematic reviews of all types

Exclusion Criteria:

* No English abstract
* Other types of evidence syntheses (e.g. scoping reviews, methodological papers)
* Protocols
* Editorials
* Others: e.g. Corrections, retractions, erratums, or summaries of SRs
* No email address available

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 1941 (Actual)
Dates: Start 2024-08-01 (Actual); Primary Completion 2024-09-30 (Actual); Study Completion 2024-09-30 (Actual)

PRIMARY OUTCOMES:
Trial participation | Immediately after reading the abstract
  The primary outcome of this RCT will be the trial participation, which is defined as the proportion of participants who read the abstract and then clicked on the "Continue" button. This will be quantified by dividing the number of participants who read the abstract and proceeded to complete the survey by the total number of individuals who clicked on the link in the email. Information will be electronically captured in SoSci survey.

SECONDARY OUTCOMES:
Indicators of a well-written abstract | Immediately after reading the abstract
  The secondary outcomes will be four indicators of a well-written abstract, as follows:
  1. Informativeness
  2. Accuracy
  3. Attractiveness
  4. Conciseness.
  The extent to which participants perceive these criteria to be fulfilled will be quantified on a 4-point Likert scale, e.g. very little informative, little informative, informative, very informative. For data analysis, the data will be dichotomized. For instance, the statements "very little informative" and "little informative" will be summarized in the category "non-informative," while the statements "informative" and "very informative" will be summarized in the category "informative."

OTHER OUTCOMES:
Time needed to read the abstract | Immediately after reading the abstract
  The time needed to read the abstract will be quantified. The time interval is defined as the period between the participant clicking on the link in the email and clicking on the "Continue" button to proceed to the survey. This time will be automatically recorded by SoSci Survey.

CONTACTS AND LOCATIONS:
Locations (1):
- Carl von Ossietzky Universität Oldenburg, Oldenburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Bahadoran Z, Mirmiran P, Kashfi K, Ghasemi A. The Principles of Biomedical Scientific Writing: Abstract and Keywords. Int J Endocrinol Metab. 2020 Jan 28;18(1):e100159. doi: 10.5812/ijem.100159. eCollection 2020 Jan. PMID 32308700
- [Background] Munn Z, Stern C, Aromataris E, Lockwood C, Jordan Z. What kind of systematic review should I conduct? A proposed typology and guidance for systematic reviewers in the medical and health sciences. BMC Med Res Methodol. 2018 Jan 10;18(1):5. doi: 10.1186/s12874-017-0468-4. PMID 29316881
- [Background] Soderberg L, Ergun O, Ding M, Parker R, Borofsky MS, Pais V, Dahm P. Percutaneous nephrolithotomy versus retrograde intrarenal surgery for treatment of renal stones in adults. Cochrane Database Syst Rev. 2023 Nov 13;11(11):CD013445. doi: 10.1002/14651858.CD013445.pub2. PMID 37955353
- [Background] Soderberg L, Ergun O, Ding M, Parker R, Borofsky M, Pais V, Dahm P. Percutaneous nephrolithotomy vs retrograde intrarenal surgery for renal stones: a Cochrane Review. BJU Int. 2024 Feb;133(2):132-140. doi: 10.1111/bju.16220. Epub 2023 Nov 29. PMID 37942649
- [Derived] Helbach J, Wandscher K, Pieper D, Hoffmann F. Readers' attention to shorter versus longer abstracts of systematic reviews: a randomised controlled trial. BMJ Evid Based Med. 2025 Oct 17:bmjebm-2024-113613. doi: 10.1136/bmjebm-2024-113613. Online ahead of print. PMID 41106849

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-07-24): https://cdn.clinicaltrials.gov/large-docs/05/NCT06525805/Prot_SAP_000.pdf